CLINICAL TRIAL: NCT00576524
Title: Application of Impedance Threshold Device Technologies to Treat and Prevent Intradialytic Hypotension in Children Undergoing Hemodialysis
Brief Title: Application of Impedance Threshold Device Technologies to Treat and Prevent Hypotension During Dialysis
Acronym: ITD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Completion not feasible. THERE ARE NO RESULTS FROM THIS TRIAL
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Advanced Circulatory Systems (Industry)
Responsible Party: Principal Investigator, Vijay Srinivasan, Attending Physician, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007-12-5712
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Results first posted 2013-02-26 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-01

CONDITIONS: Intradialytic Hypotension; End Stage Renal Disease; Low Blood Pressure
Keywords: Hypotension during dialysis; End Stage Renal Disease; Decrease complications during dialysis; Low Blood Pressure
MeSH Terms: conditions — Kidney Failure, Chronic; Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham Device first, ITD next (Experimental): Subjects will be randomized to recieve sham device first, ITD next after washout of 7 days.
  Interventions: Device: ITD; Device: Sham
- ITD first, sham device next (Experimental): Subjects will be randomized to receive ITD first, sham device next, after washout of 7 days.
  Interventions: Device: ITD; Device: Sham

INTERVENTIONS:
Device: ITD — ITD will be applied for 30 minutes at a time with 10 minute breaks for the entire duration of hemodialysis on 2 separate occasions
  Other Names: ResQpod
Device: Sham — Sham will be applied for 30 minutes at a time with 10 minute breaks for the entire duration of hemodialysis on 2 separate occasions

SUMMARY:
The purpose of this study is to evaluate the application of the impedance threshold device during hemodialysis in children to optimize fluid removal, reduce the incidence of complications (such as cramps,vomiting and hypotension), and device tolerance.

DETAILED DESCRIPTION:
Effective fluid removal during hemodialysis is one of the biggest challenges in children with end-stage renal disease (ESRD). Generally, children do not tolerate having more than 3-4% of their body weight removed during each dialysis session thus necessitating multiple sessions each week to ensure effective renal replacement. Excessive fluid removal is often associated with nausea, vomiting, hypotension and cramps resulting in serious complications in patient care during and immediately after dialysis as well as reduced patient compliance. The development of novel therapies to increase the amount of fluid removed during each session without a corresponding increase in the incidence of complications is therefore very important to improve quality and compliance with hemodialysis; and eventually survival of children with ESRD. The purpose of this study is to evaluate the application of the impedance threshold device during hemodialysis in children to optimize fluid removal, reduce the incidence of complications (such as cramps,vomiting and hypotension), and device tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 8-18 years of age
* Subjects undergoing hemodialysis for ESRD

Exclusion Criteria:

* Subjects less than 8 years old or greater than 18 years old.
* Hemodialysis for indications other than ESRD.
* Current symptoms of chest pain, shortness of breath, fever, presence of dilated cardiomyopathy, unstable congestive heart failure, pulmonary hypertension, atrial fibrillation, hyperthyroidism, and aortic stenosis.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2008-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Srinivasan, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited subjects from September 2007 to February 2011. The study will be performed in the Dialysis Unit of the Division of Nephrology, Department of Pediatrics at the Children's Hospital of Philadelphia (CHOP) with informed consent.
Pre-assignment Details: The study design will consist of a "run-in phase", followed by a randomized, cross-over, clinical "intervention phase" with application of the ITD (sham or -7 cm H2O) in 20 pediatric subjects undergoing regular hemodialysis.
Groups:
- ITD First, Sham Device Next: A group of subjects will be randomized to receive the ITD first, followed by sham 7 days later.
- Sham Device First, ITD Next: A group of subjects will be randomized to receive sham first, followed by ITD 7 days later.
Period: Overall Study
Arm/Group | ITD First, Sham Device Next | Sham Device First, ITD Next
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sham Device: A group of subjects will be randomized to receive the placebo sham device.
- ITD Device: A group of subjects will be randomized to receive Impedance Threshold Device.
- Total: Total of all reporting groups
Arm/Group | Sham Device | ITD Device | Total
Number analyzed (Participants) | 2 | 0 | 2
Age Categorical [Number; unit: participants]
  <=18 years | 2 |  | 2
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Data not analyzed- study closed due to lack of recruitment |  | 0
  Male | NA — Data not analyzed- study closed due to lack of recruitment |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Fluid Removal
Description: Fluid removed as percentage of dry body weight.
Time Frame: 6 weeks
Population: Data not analyzed - study closed due to lack of recruitment
Groups:
- Sham Device First, ITD Next: A group of subjects will be randomized to receive the sham device, followed by ITD next after 7 days.
- ITD First, Sham Device Next: A group of subjects will be randomized to receive ITD, followed by sham device after 7 days.
Arm/Group | Sham Device First, ITD Next | ITD First, Sham Device Next
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Extra Days to Achieve Target Dry Weight
Description: Extra number of days required for hemodialysis/ultrafiltration to achieve dry body weight
Time Frame: 6 weeks
Population: Data not analyzed - study closed due to lack of recruitment
Groups:
- Sham Device First, ITD Next: A group of subjects will be randomized to receive the sham device, follwed by ITD 7 days later.
- ITD First, Sham Device Next: A group of subjects will be randomized to receive ITD, followed by sham device 7 days later.
Arm/Group | Sham Device First, ITD Next | ITD First, Sham Device Next
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Changes in Heart Rate and Blood Pressure Measured by a Non-invasive Cuff.
Time Frame: 6 weeks
Population: Data not analyzed - study closed due to lack of recruitment
Arm/Group | Sham Device | ITD Device
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Sham Device | ITD Device
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes